CLINICAL TRIAL: NCT03111992
Title: Phase I/Ib, Multi-center, Open-label, Study of Single Agent CJM112, and PDR001 in Combination With LCL161 or CJM112 in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study of Single Agent CJM112, and PDR001 in Combination With LCL161 or CJM112 in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2106
Record Dates: First submitted 2017-03-22; First posted 2017-04-13 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
Keywords: Myeloma,; Multiple Myeloma,; Hematologic Diseases,; Myeloma, Multiple,; Myeloma-Multiple,; Programmed Cell Death 1 Receptor
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Hematologic Diseases | interventions — spartalizumab; LCL161

STUDY DESIGN:
Intervention Model Description: The study is comprised of 3 treatment arms:
  * Single agent CJM112 (Arm A)
  * A fixed dose of PDR001 in combination with CJM112 (Arm B)
  * A fixed dose of PDR001 in combination with LCL161 (Arm C)
  Patients may switch from treatment on Arm A to the corresponding CJM112 dose level on Arm B at the time of disease progression if that dose level has been declared safe, and if patients do not have any DLTs on single agent CJM112. Otherwise, patients will switch to a lower dose level that has been declared safe. No other cross-over between treatment arms is allowed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Dose escalation of single agent CJM112
  Interventions: Drug: CJM112
- Arm B (Experimental): Dose escalation of CJM112 in combination with a fixed dose of PDR001
  Interventions: Drug: PDR001; Drug: CJM112
- Arm C (Experimental): Dose escalation of LCL161 in combination with a fixed dose of PDR001
  Interventions: Drug: PDR001; Drug: LCL161

INTERVENTIONS:
Drug: PDR001 — Anti-PD1 antibody
  Arms: Arm B; Arm C
Drug: CJM112 — Anti-IL-17A antibody
  Arms: Arm A; Arm B
Drug: LCL161 — Oral small molecule SMAC-mimetic
  Arms: Arm C

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and identify the recommended doses of single agent CJM112, and of CJM112 or LCL161 in combination with PDR001, in patients with relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent before any screening procedures.
* Male or female patients ≥18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Patients with a confirmed diagnosis of multiple myeloma who have received two or more lines of therapy including an IMiD and PI, and are relapsed and/or refractory to their most recent line of therapy. Patients who have received a prior autologous bone marrow transplant and otherwise meet the inclusion criteria are eligible for this study.
* Must have measurable disease defined by at least 1 of the following 3 measurements:
* Serum M-protein ≥ 0.5 g/dL OR
* Urine M-protein ≥ 200 mg/24 hours OR
* Serum free light chain (FLC) > 100 mg/L of involved FLC
* All patients must be willing to undergo a mandatory serial bone marrow aspirate and/or biopsy at screening and subsequently following treatment for the assessment of biomarker/pharmacodynamics and disease status. Exceptions may be considered after documented discussion with Novartis.

Other inclusion criteria included in the protocol might apply.

Exclusion Criteria:

* Use of systemic chronic steroid therapy (≥10mg /day of prednisone or equivalent), or any immunosuppressive therapy within 7 days of first dose of study treatment. Topical, inhaled, nasal, or ophthalmic steroids are allowed.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
* Active, known or suspected autoimmune disease other than patients with vitiligo, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur.
* Patients with prior known toxicity attributed to PD-1 or PDL-1 directed therapy, which led to discontinuation of these agents, will be excluded from the PDR001 containing arms of the study.
* Patients with prior known toxicity from IL-17A directed therapy, which led to discontinuation of the study treatment, will be excluded from CJM112 containing arms of the study.
* Any of the following clinical laboratory results during screening (i.e., within 28 days before the first dose of study treatment):

  * Absolute neutrophil count (ANC) < 1,000/mm3 without growth factor support within 7 days prior to testing
  * Platelet count < 75,000 mm3 without transfusion support within 7 days prior to testing
  * Bilirubin > 1.5 times the upper limit of the normal range (ULN)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN
  * Calculated creatinine clearance < 30 ml/min according to Cockcroft-Gault equation Other exclusion criteria included in the protocol might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting dose limiting toxicities | 2 months
  number of patients reporting dose limiting toxicity
The number of patients who experience a treatment-related adverse event after being treated with a single dose of single agent CJM112, or two doses of PDR001 in combination with CJM112 or LCL161 | 24 months
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.0
The number of patients requiring interruptions after a single dose of single agent CJM112, or two doses of PDR001 in combination with CJM112 or LCL161 | 24 months
  Frequency of patients requiring a dose interruption
The number of patients treated with single agent CJM112, or PDR001 in combination with either CJM112 or LCL161, who discontinued treatment | 24 months
  Frequency of patients discontinuing treatment.
The number of patients requiring a dose reduction after a single dose of single agent CJM112, or two doses of PDR001 in combination with CJM112 or LCL161 | 24 months
  Frequency of patients requiring a dose reduction.

SECONDARY OUTCOMES:
Immunogenicity of PDR001 and CJM112 | First 6 months of study treatment
  Presence and/or concentration of anti-PDR001, and anti-CJM112 antibodies
Overall Response Rate (ORR) | 24 Months
  Determine ORR in each arm of the study
Best Overall Response (BOR) | 24 Months
  Determine BOR in each arm of the study
Progression Free Survival (PFS) | 24 Months
  Determine PFS in each arm of the study
Disease Control Rate (DCR) | 24 Months
  Determine DCR in each arm of the study
AUC of PDR001, CJM112 and LCL161 | 24 months
  AUC
Cmax of PDR001, CJM112 and LCL161 | 24 months
  Cmax
Tmax of PDR001, CJM112 and LCL161 | 24 months
  Tmax
Half-life of PDR001, CJM112 and LCL161 | 24 months
  Half-life
Concentration vs time profile of PDR001, CJM112 and LCL161 | 24 months
  Concentration vs time

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (2):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Milan, MI, Italy
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=717
- See also: Results for CPDR001X2106 can be found on the Novartis Clinical Trial Results Website. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17798